CLINICAL TRIAL: NCT05900544
Title: Maximizing Benefit of Lung Cancer Screening Incidental Findings of Cardiovascular, Respiratory and Breast Measures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded by AHRQ
Sponsor: University of Montana (Other)
Responsible Party: Principal Investigator, Curtis Noonan, Principal Investigator, University of Montana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-0592-P0001
Record Dates: First submitted 2023-05-28; First posted 2023-06-12 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Coronary Disease; Emphysema or COPD; Breast Density
MeSH Terms: conditions — Coronary Disease; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Quasi-experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implementation (Experimental): New lung cancer screening participants with clinically significant incidental findings received new patient-centered report
  Interventions: Other: System implementation of patient-centered incidental findings report

INTERVENTIONS:
Other: System implementation of patient-centered incidental findings report — For three lung cancer screening programs a system level implementation for a patient-centered incidental findings report

SUMMARY:
The investigators will implement a patient-centered outcomes tool for participants in lung cancer screening programs that receive clinically important incidental findings relevant to heart, breast and lung health. The study objective is to evaluate participant response and clinical follow-up following implementation of a patient-centered incidental findings communication tool.

DETAILED DESCRIPTION:
A computer assisted personal interview survey will be administered by study personnel to capture information about perceived risk, cues to action and self-efficacy among lung cancer screening participants. Participants eligible for recruitment will have had incidental findings from the low dose CT: moderate to severe CAC, grade 3 or 4 breast density, moderate to severe emphysema, or multiple incidental findings. The interview-administered survey will be conducted by telephone with responses entered by study personnel into a REDCap database. The REDCap questionnaire will be adapted to a given patient's IF status. The survey questions will be based on the Health Belief Model that has been used effectively in the context of secondary prevention. For each participant the survey will be conducted before and after system level implementation of a patient-centered incidental findings communication tool.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for lung cancer screening program
* Presence of one of three incidental findings on low dose CT: coronary artery calcification, extensive breast density (for females), or emphysema

Exclusion Criteria:

* No incidental findings from lung cancer screening low dose CT

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Precaution Adoption Process Model (PAPM) health behavior stage | 3 years
  The PAPM is a theoretical, stages of change model that, in conjunction with the Health Belief model, has been used to guide the study of health behaviors, including to promote screening for health conditions. The PAPM outlines seven stages along a continuum toward health behavior change: (1) unaware of the health behavior, (2) aware but unengaged with the health behavior, (3) engaged and thinking about acting (deciding), (4) decided not to act, (5) decided to act (but not yet acting), (6) acting, and (7) maintenance of the health behavior. Using a questionnaire, we will capture the participants' stage of change before and after implementation of the incidental findings communication tool. The desired directionality of change is a higher stage with 7 being the maximum score and 1 being the minimum score.